CLINICAL TRIAL: NCT00934362
Title: A Double Blind, Cross-Over Study Comparing Aerosolized Lucinactant and Vehicle on Mucociliary Clearance for Cystic Fibrosis Lung Disease
Brief Title: Effect of Lucinactant on Mucus Clearance in Cystic Fibrosis Lung Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Cystic Fibrosis Foundation (Other); Windtree Therapeutics (Industry)
Responsible Party: Principal Investigator, Scott Donaldson, MD, MD, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-0795; KL4-CF-01; DONALD04A0
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Results first posted 2013-02-20 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2013-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lucinactant; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lucinactant first, then placebo (Other): Active treatment first, then washout period, then placebo treatment
  Interventions: Drug: Lucinactant first
- Placebo treatment first, then lucinactant treatment (Other): 0.9% NaCl vehicle treatment first, then washout period, then lucinactant treatment
  Interventions: Drug: Placebo first

INTERVENTIONS:
Drug: Lucinactant first — lucinactant 120 mg (20 mg/ml) x 5 doses over 24 hours, then washout period x 14 days, then vehicle x 5 doses over 24 hrs
  Other Names: KL-4 surfactant, lucinactant, aerosurf
  Arms: Lucinactant first, then placebo
Drug: Placebo first — 6 mL normal saline x 5 doses over 24 hours, then washout period x 14 days, then lucinactant x 5 doses over 24 hours
  Other Names: normal saline; 0.9% NaCl
  Arms: Placebo treatment first, then lucinactant treatment

SUMMARY:
Mucus clearance is impaired in cystic fibrosis. Inhaled surfactants may reduce adhesive forces between mucus and airway surfaces and improve mucus clearance. This in turn my improve lung health. The investigators propose to measure mucus clearance before and after lucinactant or vehicle administration in patients with cystic fibrosis.

DETAILED DESCRIPTION:
This single-center pilot study is designed as a double-blind, randomized, cross-over clinical trial to evaluate the effects of inhaled lucinactant, an investigational peptide-containing synthetic surfactant (6 ml of 20 mg total phospholipid (TPL)/mL solution x 5 doses) in patients with mild to moderate CF lung disease. Lucinactant and vehicle will be delivered via a 510k approved vibrating mesh nebulizer, the Pari eFlowTM. The study duration corresponds to a 2-10 day screening phase, followed by a 20 day post-randomization phase that consists of two treatment periods (3 days each) and a washout period (14 days). A total of 16 patients will be enrolled and randomly assigned to one of two treatment sequences (Lucinactant followed by vehicle or vehicle followed by lucinactant). The primary outcome will be the rate of MC, as assessed via gamma scintigraphy, post-lucinactant and post vehicle. Secondary outcomes will include the rate of cough clearance (CC), lung clearance index (LCI), absolute change from baseline in FEV1 after 5 doses of study medication, CF-specific quality of life score (via CFQ-R instrument), in vitro assessments of sputum rheology, and various safety parameters.

ELIGIBILITY:
Inclusion Criteria:

* Cystic fibrosis
* FEV1>40%

Exclusion Criteria:

* Unstable lung disease
* Unable or unwilling to stop hypertonic saline and dornase alfa for 3 days prior to each study period
* Relevant drug allergy or intolerance
* Recent investigational drug use (30 days)

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott H Donaldson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: two week washout period between treatment phases of this cross-over study
Groups:
- Lucinactant First, Then Placebo: 20 mg/ml x 6 ml (5 doses) lucinactant then 0.9% NaCl x 6 ml (5 doses)
- Placebo First, Then Lucinactant: 0.9% NaCl x 6 ml (5 doses) then 20 mg/ml x 6 ml lucinactant (5 doses)
Period: Overall Study
Arm/Group | Lucinactant First, Then Placebo | Placebo First, Then Lucinactant
Started | 8 | 8
Completed | 7 | 8
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lucinactant First, Then Placebo | Placebo First, Then Lucinactant | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (8.8) | 25.9 (6.4) | 27.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16
Baseline Mucociliary Clearance Rate [Mean (Standard Deviation); unit: Percentage Clearance] — Radiolabeled particle clearance through 60 minutes (post inhalation) is averaged as index of clearance.
  Percentage Clearance | 9.2 (4.8) | 12.0 (10.5) | 10.5 (8.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mucociliary Clearance
Description: Clearance of radiolabeled particles, following inhalation, are followed over time. Average clearance rate through 60 minutes post inhaled isotope deposition is calculated. Absolute difference between baseline and post-treatment (e.g. <60 minutes after the last dose of lucinactant or placebo) reported.
Time Frame: 1 hour after final treatment (5th dose) minus baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percent clearance
Groups:
- Lucinactant: 20 mg/ml x 6 ml lucinactant (5 doses)
- Placebo: 0.9% NaCl x 6 ml (5 doses)
Arm/Group | Lucinactant | Placebo
Number analyzed (Participants) | 15 | 15
percent clearance | 7.4 (9.3) | 9.5 (10.0)

2. Secondary Outcome: Spirometry
Description: Percent change (relative) in FEV1 between pre-treatment baseline and following 5 doses of study treatment. Post treatment values obtained 3 and approximately 22 hours after 5th dose were averaged to determine the treatment effect.
Time Frame: after 5 doses
Population: per protocol
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Lucinactant | Placebo
Number analyzed (Participants) | 15 | 15
percent change | .81 (.9) | .23 (1.1)

ADVERSE EVENTS:
Groups:
- Lucinactant: 20 mg/ml x 6 ml (5 doses)
Arm/Group | Lucinactant | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 6/16 | 8/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lucinactant (N=16) | Placebo (N=15)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
sinonasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
headache (Nervous system disorders) | 1 (1) | 2 (2)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1)
Decreased lung function (Investigations) | 1 (1) | 0 (0) — FEV1 measured after first dose of study medication
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cystic Fibrosis exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less